CLINICAL TRIAL: NCT06148610
Title: Evaluation of the Impact of the Use of the Digital Solution NewSpringForMe on Transplanted Patients' Quality of Life and Support (Bone Marrow or Peripheral Stem Cells Allotransplantation)
Brief Title: Evaluation of the Impact of the Use of NewSpringForMe on Transplanted Patients' Quality of Life and Support
Acronym: NSFM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fonds de Dotation HTC Project (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other); Nutricia Nutrition Clinique (Industry); Clinicprosport (Unknown); ELLYE (Unknown); Association Aïda (Unknown); Gilead Sciences (Industry); Pfizer (Industry); Groupe Apicil (Unknown); Association Laurette Fugain (Unknown); Fondation du LEEM (Unknown); Fondation AFNIC (Unknown); Pierre Fabre Medicament (Industry); Novartis Pharmaceuticals (Industry); University Hospital, Clermont-Ferrand (Other); LAPSCO, Université Clermont-Auvergne (Unknown)
Responsible Party: Sponsor
Other Study IDs: HTC-NSFM-121; 2021-A03034-37 (Other: Comité de Protection des Personnes Ouest IV)
Record Dates: First submitted 2023-09-07; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hematologic Diseases; Bone Marrow Transplantation; Hematopoietic Stem Cell Transplantation
Keywords: Digital solution; Companion; Quality of life; Support; Hematopoietic Stem Cell Transplantation; Post-transplant complications; Psychological, physical and nutritional balance maintenance; Bone marrow Transplantation
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NewSpringForMe cohort: Patients with hematological diseases intended to be allotransplanted (bone marrow or Hematopoietic Stem Cells)
  Interventions: Device: NewSpringForMe digital solution

INTERVENTIONS:
Device: NewSpringForMe digital solution — Follow-up of transplanted patients for hematological diseases using the NewSpringForMe device as support of quality of life

SUMMARY:
Bone marrow transplantation is both a great treatment for patients with hematological diseases. It is also one of the only hopes of staying alive by "starting from scratch". It is a trying life experience, at all its stages. To support these patients and increase their success in healing and returning to a "normal life", quality of life is an ally of choice for the success of care.

NewSpringForMe is an innovative tool designed for the benefit of transplant patients, through the deployment of unprecedented interdisciplinary support benefiting from the best digital technologies. This digital solution is aimed at all patients, adults and pediatrics, before, during and after bone marrow transplantation, in a long-term approach. NewSpringForMe results from the multidisciplinary collaboration of medical and paramedical experts in the field of hematology and transplantation, as well as in the field of psychology.

With NewSpringForMe, each transplant patient has a personalized and scalable space accessible via a web platform, constantly offering, according to their needs and at their own pace, a range of recommendations, tools and exercises in psychology, nutrition / dietetics and physical activity, the three pillars of overall well-being. Perfectly integrated into the care pathway and the transplant protocol, from the announcement of the treatment to the long-term follow-up, several years after the intervention, NewSpringForMe complements the medical treatments provided by the medical profession: the communication of the assessments from the platform as well as patient data for caregivers allows adaptation of therapies and optimization of medical care. Thanks to the consideration of individual parameters and their evolution, and thanks to specific algorithms, each tool is adapted to the course of care and to the life of each patient, as well as to their personal health situation throughout their transplant journey.

In order to demonstrate the benefits of using NewSpringForMe, the project plans to evaluate the platform and its impact on the quality of life in patients with hematological diseases. This evaluation will be done by the patients themselves and by the nursing staff. The evaluation will be carried out using a monocentric approach on a pilot cohort. The objective is to demonstrate that integrative health ensuring simultaneous care of body and mind increases the chances of success of the transplant while limiting post-transplant complications.

DETAILED DESCRIPTION:
Each year in France, nearly 2,000 patients, adults and children of all ages, are treated by bone marrow transplantation, the last therapeutic resort to treat and cure serious blood diseases, malignant or not. If this intervention saves more and more lives, it can lead to early or late complications in 50% of patients (graft versus host disease or GvHD in English for Graft versus Host Disease, cardiac and/or metabolic complications, etc.), very disabling on a daily basis and fatal in 25% of cases. The chances of success of the bone marrow transplant are directly correlated to the non-occurrence of these complications.

A mutual influence of psychological health and physical health on the chances of success of the transplant has been highlighted for several years. Simultaneous support of the mind and body based on the 3 pillars - nutritional, psychological, physical - would ensure better preparation for the transplant process for faster recovery after it thanks to the limitation of the occurrence of complications.

However, to date there is no comprehensive support program covering both mental and physical health to help patients overcome the difficulties associated with the transplant and the return to social and professional life.

As part of their care pathway, patients can benefit from sectorized support but it remains incompletely developed, which can generate in patients a feeling of abandonment on the part of the medical team once the cancer treatment is complete.

It is in this context that the digital support solution for transplant patients, called NewSpringForMe, emerged. This project is on the initiative of Professor Régis Peffault de Latour, hematologist-transplanter at Saint-Louis Hospital in Paris. The latter relied on more than 15 years of experience in contact with transplant patients to highlight an unmet need in terms of support. This need is for therapeutic support that complements care, reinforcing it, and making each patient the main actor in his or her quality of life. To fill this gap, the interdisciplinary support tool, NewSpringForMe, combining psychology, nutrition and adapted physical activity, was developed. Thanks to a global management of these three dimensions throughout the transplant process (in the hospital but also in his daily life), NewSpringForMe aims at a better preparation and a more global management of the patient, condition of the best live towards his remission, by making him actor of his course of care.

NewSpringForMe is the first global support system developed in the field of bone marrow transplantation by an entity independent of healthcare structures, thus giving the tool greater accessibility to patients regardless of their prescribing hospital structure.

The innovation of the project is based on comprehensive support for bone marrow transplant patients in three dimensions: psychology, nutrition and physical activity, with the NewSpringForMe digital tool.

Designed around interconnected spaces, NewSpringForMe offers each patient, permanently, according to their needs and at their own pace, a range of tools and therapeutic exercises, complementary to the care provided by the medical and nursing profession, depending on their condition. progress in the transplant process.

* Nature: web platform providing more versatility, flexibility and maneuverability
* Transversality: integrative health for optimized preparation and comprehensive support
* Integration into the care pathway for long-term follow-up

A public health approach: NewSpringForMe's challenge is not only to improve support for patients, but also to keep them healthy throughout their bone marrow transplant experience, thus being part of a optimization of the French healthcare system for better social and professional reintegration.

A therapeutic tool, a place of exchange and sharing, a facilitator of social ties: success is based on the creation of a real dynamic of community of patients and on the increase of knowledge, in order to improve their care.

In order to measure the impact of the use of the NewSpringForMe digital solution, a monocentric pilot phase of evaluation is planned in a cohort of 150 to 200 patients allografted by bone marrow within the hematology transplant department of the Hospital Saint-Louis de Paris (AP-HP).

Recruitment: The NewSpringForMe support solution will be offered directly by the healthcare team (transplant doctor, transplant coordinator, etc.) to the patient identified to benefit from a transplant protocol and who meets the inclusion/exclusion criteria above. The medical team will submit the consent and information leaflet to the patient likely to be included. This protocol will be presented and carried out, if accepted by the patient, as part of routine care. Each patient included must provide written informed consent.

The impact study provides for a longitudinal follow-up of the patients included, based on their transplant journey. A follow-up of 1 year from the inclusion of the patient to the announcement of the transplant will make it possible to assess in a relevant way the impact of the use of the platform, to identify medium-term profiles in relation to the events post-transplant (relapse, complications, etc.). The duration of the project, including inclusion and follow-up of patients, analysis and exploitation of results, is estimated at 24 months.

To date, the IT development of the platform is 85% complete; improvements still need to be made to optimize the tool, the generation and the collection of data. In addition, the enrichment of the platform continues with the integration of visually optimized illustrations and cooking recipes adapted to diets in the journey of the transplant patient.

Once the impact has been demonstrated and assuming positive results, the digital solution can be deployed on a national scale, in all French allograft centers. This deployment will be carried out in collaboration with the Francophone Society of Bone Marrow Transplantation and Cellular Therapy (SFGM-TC) and the Biomedicine Agency. It will be aimed at all transplant patients for a serious cancerous blood disease - leukemia, lymphoma, etc. - or not, adults and pediatrics, representing a population of approximately 2,000 people per year (see annual activity reports of the Biomedicine Agency). Given the growing number of patients going for transplant, the development and implementation of this support program will have a strong impact in the medico-social field. These arguments also support the long-term viability of this support program.

ELIGIBILITY:
Inclusion criteria :

* at least 18 years old
* with a first indication for allograft bone marrow or Peripheric Stem Cells
* monitored by the adult hematology transplant department St-Louis Hospital
* having signed the consent
* affiliated to a social security scheme
* able to understand the objectives of the study and to use a digital tool

Exclusion criteria :

* aged under 18
* with an indication of second or third allograft
* not being affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with haemopathies, malignant or not, justifying a first indication of bone marrow or peripheral stem cells allo transplantation
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative affects | 12 months
  Level of negative affect (PHQ, Patient Health Questionnaire, Spitzer et al., 2006). Scales measuring sad mood in 9 items (from 0 "never" to 3 "almost every day") and anxious mood in 7 items (from 0 "never" to 3 "almost every day").
  Simple Verbal Scale (EVS) for assessing pain intensity (from 0 "no pain" to 10 "maximum pain imaginable").
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Positive affects | 12 months
  Level of positive affects (SA-DHS, Subjective Authentic Durable Happiness Scale, Dambrun et al., 2012). Scale of 13 items (from 1 "very low" to 7 "very high") measuring the level of well-being.
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Life quality | 12 months
  Quality of life (SF-12, Gandek, Ware & Aronson, 1998)
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Life values | 12 months
  Identification of life values (Valued Living Questionnaire, Wilson & Groom, 2002). 10-item scale (from 1 "not at all important" to 10 "very important").
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Mindfulness | 12 months
  Level of dispositional mindfulness (FFMQ-15, 15 item Five Facets Mindfulness Questionnaire, Baer et al., 2008; Gu et al., 2016) in 15 items (from 1 "never true" to 5 "always true")
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Pain intensity | 12 months
  Simple Verbal Scale (EVS) for assessing pain intensity (from 0 "no pain" to 10 "maximum pain imaginable")
  Data will be collected at each connection and each time the platform and spaces used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Physical effort | 12 months
  Stress test: TM6 walking test (distance in meters measured for 6 minutes)
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Physical suppleness | 12 months
  Shoulder flexibility test and lower limb spine test (in centimeters). For the shoulder test, the distance is calculated between the two hands located behind the back of the individual performing the test. For the lower limb spine test, the distance measured is the finger-to-ground distance.
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Physical activity level | 12 months
  Level of physical activity using a specific self-assessment questionnaire (see J. Ricci and L. Gagnon, University of Montreal, modified by F. Laureyns and JM. Séné) to measure physical activity and determine a profile (inactive, active, very active) depending on the score (ranging from 0 to 5).
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Fatigue | 12 months
  Fatigue assessed by the Pichot scale (see "Scales and assessment tools in general medicine" J. Gardenas et Coll. -Le Généraliste- Supplement to No. 2187; March 2002). This scale allows you to calculate the level of fatigue (from 0 not at all to 4 extremely). It includes 8 items: "I lack energy", "everything requires effort", "I feel weak in certain parts of the body", "my arms or legs are heavy", "I feel tired without reason", "I want to lie down to rest", "I have difficulty concentrating", "I feel tired, heavy and stiff".
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Body mass index | 12 months
  Function of the weight in kg and the height in m
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Appetite quality | 12 months
  Using a scale
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment
Ingested quantities | 12 months
  Food intake using the food intake assessment tool (EPA).
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Eating disorders | 12 months
  Occurrence of eating disorders such as nausea, vomiting, inappetence, dysgesia, dysphagia
  Data will be collected at each connection and each time the platform and spaces are used. However, a connection to the platform and to the psychology, nutrition and physical activity spaces will be required at times defined as follows, in order to allow data collection on basic times applicable to all patients and to allow a relevant assessment.
Occurrence and extent of post-transplant complications and post-transplant recovery | 12 months
  * Nature, frequency of occurrence and extent of post-transplant complications.
  * Number of therapeutic protocols initiated to treat complications
  These data relating to post-transplant complications will not be collected from the NewSpringForMe platform but collected from the patient's medical file by the team caregiver.
  All these outcomes will be aggregated to achieve a final score related to the post-transplant complications
Occurrence of hospitalizations | 12 months
  - Average cumulative duration (in days) of unscheduled hospitalizations
  These data relating to post-transplant complications will not be collected from the NewSpringForMe platform but collected from the patient's medical file by the team caregiver.
Post-transplant recovery | 12 months
  * Overall survival
  * Occurrence of relapse
  * Recovery
  These data relating to post-transplant complications will not be collected from the NewSpringForMe platform but collected from the patient's medical file by the team caregiver. They will be aggregated to arrive to a final score combining their values.

SECONDARY OUTCOMES:
Admissibility of NewSpringForMe and its tools in terms of attractiveness, understanding, usefulness and relevance | 12 months
  * Number of connections to the platform
  * Overall duration of use of the platform and by space
  * Perceived ease of use (e.g. accessibility, ergonomics), perceived usefulness, positive and negative attitude towards the tool (appreciation of content, functionality), intention to use
  All these outcomes will be assessed by scales that share common unit measure. They will be aggregated to achieve a radar graph.

CONTACTS AND LOCATIONS:
Overall Officials: Régis Peffault de Latour, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service Hématologie Greffe Trèfle 3, Hôpital Saint-Louis, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
Would depend on the results obtained from the pilot study

REFERENCES:
- [Background] Dirou S, Chambellan A, Chevallier P, Germaud P, Lamirault G, Gourraud PA, Perrot B, Delasalle B, Forestier B, Guillaume T, Peterlin P, Garnier A, Magnan A, Blanc FX, Lemarchand P. Deconditioning, fatigue and impaired quality of life in long-term survivors after allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2018 Mar;53(3):281-290. doi: 10.1038/s41409-017-0057-5. Epub 2017 Dec 21. PMID 29269801
- [Background] Brotelle T, Lemal R, Cabrespine A, Combal C, Hermet E, Ravinet A, Bay JO, Bouteloup C. Prevalence of malnutrition in adult patients previously treated with allogeneic hematopoietic stem-cell transplantation. Clin Nutr. 2018 Apr;37(2):739-745. doi: 10.1016/j.clnu.2017.03.016. Epub 2017 Mar 28. PMID 28390845
- [Background] Corman M, Rubio MT, Cabrespine A, Brindel I, Bay JO, Peffault De La Tour R, Dambrun M. Mental health and quality of life of patients undergoing hematopoietic stem cell transplantation (HSCT) prior to hospitalization: a cross-sectional complete state health study. Health Psychol Behav Med. 2021 Jan 28;9(1):70-83. doi: 10.1080/21642850.2021.1873140. PMID 34104550
- [Background] Hoodin F, Uberti JP, Lynch TJ, Steele P, Ratanatharathorn V. Do negative or positive emotions differentially impact mortality after adult stem cell transplant? Bone Marrow Transplant. 2006 Aug;38(4):255-64. doi: 10.1038/sj.bmt.1705419. Epub 2006 Jun 19. PMID 16785869
- [Background] Kisch A, Lenhoff S, Zdravkovic S, Bolmsjo I. Factors associated with changes in quality of life in patients undergoing allogeneic haematopoietic stem cell transplantation. Eur J Cancer Care (Engl). 2012 Nov;21(6):735-46. doi: 10.1111/j.1365-2354.2012.01354.x. Epub 2012 Apr 23. PMID 22519415
- [Background] Snowden JA, Sanchez-Ortega I, Corbacioglu S, Basak GW, Chabannon C, de la Camara R, Dolstra H, Duarte RF, Glass B, Greco R, Lankester AC, Mohty M, Neven B, de Latour RP, Pedrazzoli P, Peric Z, Yakoub-Agha I, Sureda A, Kroger N; European Society for Blood and Marrow Transplantation (EBMT). Indications for haematopoietic cell transplantation for haematological diseases, solid tumours and immune disorders: current practice in Europe, 2022. Bone Marrow Transplant. 2022 Aug;57(8):1217-1239. doi: 10.1038/s41409-022-01691-w. Epub 2022 May 19. PMID 35589997
- See also: Description of NewSpringForMe digital solution — https://www.htcproject.org/projet/newspringforme/